CLINICAL TRIAL: NCT05934994
Title: Contribution of MUltiparametric Analysis in Bone Scintigraphy for the Characterisation of Solitary Bone Lesions Whose Malignant Origin Cannot be Excluded on Conventional Imaging
Brief Title: Contribution of MUltiparametric Analysis in Bone Scintigraphy for the Characterisation of Solitary Bone Lesions
Acronym: MUSIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Achraf BAHLOUL, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022PI051
Record Dates: First submitted 2023-03-28; First posted 2023-07-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Bone Lesion

STUDY DESIGN:
Intervention Model Description: People with indeterminate solitary bone lesions on conventional imaging, for whom a biopsy or surgery is scheduled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with undetermined solitary bone lesions (Experimental): All patients with indeterminate solitary bone lesions undetermined on conventional imaging for whom a biopsy or excision is scheduled, will be able to participate in the study.
  Interventions: Other: Bone scan

INTERVENTIONS:
Other: Bone scan — the bone scintigraphy will include 3 stages: study of perfusion then early tissue uptake and finally late bone fixation
  Other Names: Bone scan in single photon emission computed tomography

SUMMARY:
The hypothesis of the study is that non-invasive Single photon emission computed tomography (SPECT-CT) bone scintigraphy makes it possible to better characterize solitary bone lesions, in particular the exclusion of their malignancy in order to avoid unnecessary biopsy and possible complications for the patient.

DETAILED DESCRIPTION:
Bone scintigraphy includes 3 stages: study of perfusion then of early tissue uptake and finally of late bone fixation.

Hyperactivity of malignant bone lesions at the 3 stages of bone scintigraphy has been reported, but on planar scintigraphic images not allowing precise anatomical localization of the lesions.

Currently, the generalization of SPECT-CT (Single Photon Emission Computed Tomography) combined with Tomodensitometry) acquisition thanks to the deployment of semiconductor cameras, makes it possible to carry out a multiparametric analysis of bone lesions with quantification of the intensity of the signal expressed in SUVmax (Standard Uptake Value maximum) at the 3 times of the scintigraphy

ELIGIBILITY:
Inclusion Criteria:

* Person, having received complete information on the organization of the research and having signed the informed consent and:

  * Age ≥ 18 years old.
  * Having read and understood the information document.
  * Affiliated to a social security scheme.
* Patient with an indeterminate solitary bone lesion on conventional imaging, for which an indication for biopsy +/- excision is planned.

Exclusion Criteria:

* Pregnant woman or woman of childbearing age and without contraceptive means or nursing mother.
* Unstable medical condition and/or inability to remain still during recordings.
* Known allergy to one of the components of the radiopharmaceutical technetium-99m-Technescan HDP (product required to perform the bone scan).
* Person referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code.
* Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care under articles L. 3212-1, L. 3213-1

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Assess the diagnostic performance of the Time To Peak parameter | 24 hours
  Sensitivity, specificity, positive predictive value and negative predictive value of the dynamic parameter Time-to-peak to characterize a benign lesion. The Time-To-Peak is defined by the time to reach the SUVmax peak, i.e. the top of the perfusion curve. The benign character is defined by criteria of biopathology at the biopsy +/- surgery.

SECONDARY OUTCOMES:
To evaluate the diagnostic performance of the Standard Uptake Value max at the early stage (2nd stage) in bone scintigraphy in the evaluation of the benign nature of indeterminate solitary bone lesions on conventional imaging. | 24 hours
  Sensitivity, specificity, Positive Predictive Value and Negative Predictive Value of the Standard Uptake Value max at the early time to characterize a benign lesion.
o evaluate the diagnostic performance of the Standard Uptake Value max at the early stage (3 rd stage) in bone scintigraphy in the evaluation of the benign nature of indeterminate solitary bone lesions on conventional imaging. | 24 hours
  Sensitivity, specificity, Positive Predictive Value and Negative Predictive Value of the Standard Uptake Value max at the late stage to characterize a benign lesion.
Evaluate the impact of multiparametric analysis (combination of Time-To-Peak, Standard Uptake Value max early and late) in the classification of solitary bone lesions in bone scintigraphy. | 24 hours
  Number of patients with a benign lesion on multiparametric bone scintigraphy analysis among patients with an indeterminate bone lesion on conventional imaging and having undergone a biopsy +/- excision, defined as: 1/ [% of benign lesions detected with multiparametric analysis in bone scintigraphy].

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France